CLINICAL TRIAL: NCT03732911
Title: Developmental Monitoring and Language Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Manuel E. Jimenez, MD, MS, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2018001244
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-06

CONDITIONS: Child Development
Keywords: Child Development; Cognitive Home Environment; Literacy promotion; Text Messages
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention arm
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will receive the following intervention bundle (1) educational materials about child development and developmental monitoring checklists; (2) age and language appropriate picture books; and (3) two tailored text messages per week for a 6-month period.

SUMMARY:
The goal of this study is to pilot test an intervention developed to enhance parent knowledge regarding child development and encourage parents to engage in activities that promote language acquisition.

DETAILED DESCRIPTION:
Our specific aim for this proposal is to pilot test an intervention developed to enhance parent knowledge regarding child development and the home cognitive environment comprised of distribution of (1) publicly available developmental monitoring materials, (2) age and language appropriate children's books, and (3) text message reminders. Participants in this intervention will receive: (1) educational materials about child development and developmental monitoring checklists; (2) age and language appropriate picture books; and (3) two text messages per week for a 6-month period. Differences in pre- and post-intervention knowledge regarding child development and the home cognitive environment will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Preferred language either English or Spanish,
2. Parent or legal guardian,
3. Age ≥ 18 years,
4. Willing to accept text messages
5. Child ≤ 20 months old

Exclusion Criteria:

1. Individuals unable to provide consent
2. Individuals who do not meet inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of child development | Visit 2 (6 months)
  We will ask parents to respond to questions regarding child development upon enrollment and at 6-month follow-up.Knowledge questions are based on CDC materials and evidence based screening tools.

SECONDARY OUTCOMES:
Home cognitive environment: | Visit 2 (6 months)
  The StimQ2 is a validated, parent-report measure of the cognitive home environment for children that assesses 4 domains: (1) availability of learning materials, (2) reading, (3) parent involvement in developmental advancement, and (4) parental verbal responsiveness. We will administer the Reading and Parental Verbal Response Scale. Participants will be asked to complete the StimQ2 pre- and post-intervention.
Frequency Shared Reading: | Visit 2 (6 months)
  To measure how often parents read to their children, they will be asked to respond to the following question at enrollment and at 6-month follow-up, "How often did you read to your child in the last week?"

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States